CLINICAL TRIAL: NCT03091764
Title: Psychometric Evaluation of a Patient-Reported Symptom Index for Non-Muscle Invasive Bladder Cancer: Field Testing
Brief Title: Evaluation of a Patient-Reported Symptom Index for NMIBC
Status: Completed | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Cancer Australia (Other); Cancer Council New South Wales (Other)
Responsible Party: Sponsor
Other Study IDs: APP1103036
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Superficial Bladder Cancer
Keywords: NMIBC; non-muscle invasive bladder cancer; Patient reported outcome; Symptom burden; Questionnaire
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NMIBC Patient High Risk: Any of the following:
  * T1 tumours
  * CIS (carcinoma in situ)
  * Multiple and recurring and large (>3cm) Ta, G1, G2 tumours (all these conditions must be presented)
  (Patients requiring intravesical Bacillus Calmette-Guérin (BCG) (immunotherapy), which starts with 6 week induction treatment and continues with maintenance for 1 to 3 years)
- NMIBC Patient Intermediate Risk: All cases between High and Low Risk
  (Patients requiring intravesical therapy which lasts between 6 weeks to 3 years)
- NMIBC Patient Low Risk: Primary, solitary, Ta, LG/G1, <3cm, no CIS
  (Patients receiving frequent cystoscopies, possible tumour resections and single instillations of postoperative chemotherapy)

SUMMARY:
This project will develop and evaluate a patient-reported symptom index to assess the impact of treatment for non-muscle invasive bladder cancer on patient burden, toxicity, symptoms and side effects. The symptom index will provide a method for assessing treatments from the patient's perspective; help healthcare professionals make better informed treatment decisions, and provide a method to be able to effectively evaluate treatments for non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
The overarching aim of this research is to develop and evaluate a patient-reported Symptom Index (SI) for individuals with NMIBC (the NMIBC-SI) that is acceptable to patients, reliable, valid and responsive, and fit for purpose in clinical trials and clinical practice.

Specific clinical aims:

* Assess and compare key Patient-Reported Outcomes (PROs) across the full range of contemporary treatments for NMIBC, and over the disease trajectory including acute treatment and 1year survivorship;
* Compare PROs between patients with low, intermediate, and high risk NMIBC.

In field test 1, 200 participants will complete one questionnaire either in hard copy (pencil and paper) or online, at a time that is convenient for the participant. The questionnaire may take up to 20 minutes to complete.

In field test 2, 250 participants will complete quality of life questionnaires at four different time points; 1) before tumour resection, 2) 1 week after resection, 3) 8 weeks after resection, and 4) 1 year after resection. The questionnaires can be completed in the clinic or at home, either in hard copy (pencil and paper) or online, at a time that is convenient for the participant but still within the relevant time point. The questionnaires may take up to 30 minutes to complete.

ELIGIBILITY:
Field test 1:

Inclusion Criteria:

* diagnosed NMIBC
* Adult (>18yrs)
* able to read and understand English
* undergoing active treatment (i.e. one week after tumour resection or intravesical therapy) or completed final treatment for NMIBC within the last week

Exclusion Criteria:

* unconscious or confused
* have cognitive impairment
* unable to speak, read and/or write in English
* diagnosed with muscle invasive disease
* unable to provide informed consent

Field test 2:

Inclusion Criteria:

* newly diagnosed NMIBC
* Adult (>18yrs)
* able to read and understand English
* after imaging or flexible cystoscopy, and before active treatment
* either before endoscopic resection, or more than 4 weeks since endoscopic resection, but before active/ongoing treatment

Exclusion Criteria:

* unconscious or confused
* have cognitive impairment
* unable to speak, read and/or write in English
* diagnosed with muscle invasive disease
* unable to provide informed consent
* currently undergoing active treatment for any bladder cancer, or finished treatment within last 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥18 years) from participating centres diagnosed with NMIBC, able to read and understand English, and give their written informed consent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
NMIBC-SI development and validation | Field test 1: once only (cross-sectional). Field test 2: baseline to post-treatment (longitudinal)
  non-muscle invasive bladder cancer symptom index (questionnaire being developed and evaluated in this study)

SECONDARY OUTCOMES:
QLQC-30 | Field test 2: four time-points over 1 year
  EORTC cancer quality of life questionnaire
NMIBC24 | Field test 2: four time-points over 1 year
  EORTC superficial bladder cancer questionnaire
NMIBC-SI long term | Field test 2: four time-points over 1 year
  non-muscle invasive bladder cancer symptom index (long-term follow-up, and differences between groups)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Patel, MBBS,PhD, Principal Investigator — University of Sydney
Locations (19):
- United States (3):
  - University of Kansas, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
- Australia (12):
  - Concord Hospital, Concord, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - The Urological Cancer Centre, Westmead Specialist Centre, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Monash Health, Moorabbin, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- University of British Columbia, Vancouver, British Columbia, Canada
- New Zealand (2):
  - Canterbury Urology Research Trust, Christchurch
  - Tauranga Urology Research, Tauranga
- Salford Royal NHS Foundation Trust, Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutherford C, King MT, Smith DP, Costa DS, Tait MA, Patel MI; NMIBC-SI Working Group. Psychometric Evaluation of a Patient-Reported Symptom Index for Nonmuscle Invasive Bladder Cancer: Field Testing Protocol. JMIR Res Protoc. 2017 Nov 8;6(11):e216. doi: 10.2196/resprot.8761. PMID 29117930